CLINICAL TRIAL: NCT03279835
Title: Evaluation of a Short Version Computerized Test for Processing Speed to Detect Cognitive Disorders in HIV+ Patients
Acronym: NEURACog
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 16-PP-09
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: HIV-1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Absence of cognitive disorder
  Interventions: Other: Classic evaluation of neurocognitive functions; Other: New evaluation of neurocognitive functions
- Asymptomatic cognitive disorder
  Interventions: Other: Classic evaluation of neurocognitive functions; Other: New evaluation of neurocognitive functions
- Symptomatic cognitive impairment
  Interventions: Other: Classic evaluation of neurocognitive functions; Other: New evaluation of neurocognitive functions
- HIV associated dementia
  Interventions: Other: Classic evaluation of neurocognitive functions; Other: New evaluation of neurocognitive functions

INTERVENTIONS:
Other: Classic evaluation of neurocognitive functions — Symbol Digit Modalities Test (SDMT)
Other: New evaluation of neurocognitive functions — Cognitive Speed Computerized Test (CSCT)

SUMMARY:
The objective of this prospective study is to evaluate the prevalence of neurocognitive impairments in HIV infected patients comparing patients with and without HAART. Recent studies have demonstrated a specific HIV infected patients neurocognitive disorders profile. These cognitive disorders concern primarily information processing speed, memory recall, attentional abilities, work related memory, executive functions, and psychometrical speed. This cognitive profile is similar to another highly documented one, described for another central nervous system disease (CNS): multiple sclerosis. In both CNS diseases, the earliest and most severe disorder is the one related to the information processing speed. For the multiple sclerosis patients, a short cognitive test (SDMT) is actually used not only to identify cognitive disorders presence, but also in order to predict a long term disability worsening. A digital version of this test (CSCT), has recently been developed in order to make this early evaluation easier. We hypothesize that CSCT alteration would also predict HAND, in HIV infected patients. A complete neuropsychological assessment is highly time and personal consuming. This short (approximatively 2 minutes) digital test would be highly helpful to identify patients, who will need a more extensive neuropsychological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV-1
* Patients followed in outpatient service, over 18 years of age

Exclusion Criteria:

* Patients infected with HIV-2
* Patients with difficulty understanding the French language
* Patients present with progressive opportunistic infection
* Patients for whom a change of psychotropic treatment was performed in the last 3 weeks
* Patients with drug and / or alcohol addiction
* Patients with a history of psychiatric disorder
* Patients with stroke, endocarditis or meningoencephalitis with severe neurological sequelae

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients infected with HIV-1
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Cognitive Speed Computerized Test (CSCT) score | at patient inclusion
  allows the evaluation of the speed of the processing of the information
Montreal Cognitive Assessment (MoCA) Score | at patient inclusion
  allows the evaluation of the overall cognitive functioning

SECONDARY OUTCOMES:
Paced Auditory Serial Addition Test (PASAT) score | at patient inclusion
  allows to evaluate the concentration capacity
Numeric Memory (WAIS-III location and back) | at patient inclusion
  short-term memory evaluation and verbal working memory
Score RL-RI16 | at patient inclusion
  allows the evaluation of episodic and long-term verbal memory
Rey figure | at patient inclusion
  allows the evaluation of the long-term capacities of visio-construction (wealth score) and planning
TMTB - TMTA Time Score | at patient inclusion
  Assessment of Mental Flexibility
Verbal fluency test | at patient inclusion
  allows the evaluation of the verbal initiation and verbal language capacities
IADL score | at patient inclusion
  allows to evaluate the symptomatic character of the disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pasteur 2 - Service de Neurologie, Nice, France